CLINICAL TRIAL: NCT01938976
Title: Efficacy of School-Based, Peer-Led Asthma and Smoking Prevention Program on CO1 Levels, Nicotine Dependence, and Smoking Behavior Among Early Adolescents in Jordan
Brief Title: Efficacy of School-Based, Peer-Led Asthma and Smoking Prevention Program on CO1 Levels and Smoking Behavior Among Early Adolescents in Jordan
Acronym: TAJPlus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Technology, Sydney (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Dr. NIHAYA AL-SHEYAB, Assistant Professor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 96/2012
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Asthma; Tobacco; Waterpipe; Cigarettes
Keywords: Asthma; Tobacco; Waterpipe; Cigarettes; Adolescents; Peer education; Jordan
MeSH Terms: conditions — Asthma; Water Pipe Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adolescent Asthma Action (Experimental): Adolescent Asthma Action in Jordan (TAJ) Plus the added class smoke free pledge will be implemented in high schools in Jordan and will be compared to the TAJ alone for its efficacy in decreasing smoking rates, lowering CO1 levela and nicotine dependence.
  Interventions: Behavioral: TAJ Plus (Adolescent Asthma Action in Jordan) Plus the added class smoke free pledge
- TAJ (Experimental): TAJ Plus the class smoke free pledge will be implemented in high schools in Jordan and compared to TAJ alone
  Interventions: Behavioral: TAJ Plus (Adolescent Asthma Action in Jordan) Plus the added class smoke free pledge

INTERVENTIONS:
Behavioral: TAJ Plus (Adolescent Asthma Action in Jordan) Plus the added class smoke free pledge — Its is a school-based peer-led asthma and smoking prevention program that aims at improving asthma control and lowering nicotine dependence among smokers.
  Other Names: Triple A in Jordan (TAJ)

SUMMARY:
Study Hypotheses:

1. adolescents in intervention schools who are given Triple A program plus ASP will show more awareness in regards to cigarettee smoking health effects and less nicotine dependencethan those in the control schools who are given Triple A alone.
2. adolescents with asthma in intervention schools who are given Triple A program plus ASP will show less asthma symptoms and better control than those in the control schools who are given Triple A alone.
3. adolescent smokers and passive smokers will exhibit higher levels of carbon monoxide (CO) in their breath than those who are not active or passive smokers.
4. there is a positive correlation between self-report questions regarding student smoking status and levels of CO in their breath

ELIGIBILITY:
Inclusion Criteria: students in grades 7 and 8 in Irbid city high schools, can speak and read in both Arabic and English, obtain parental agreement, attend regular school.

-

Exclusion Criteria:students with other chronic diseases (rather than asthma),

-

Ages: 11 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 815 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
nicotine dependence level | 3 months
  Self-administered nicotine dependence scale will be used in order to measure nicotine dependence level for adolescent smokers and passive smokers
Asthma Contol level | 3 months
  The pictorial version of the asthma control test will be measured for adolescents with asthma and recent wheezing

SECONDARY OUTCOMES:
Carbon monoxide (CO) breath test | 3 months
  CO levels will be tested in adolescents' breath
knowledge about health effects of cigarettee smoking | 3 months